CLINICAL TRIAL: NCT03951389
Title: INST 1204: PIK3CA Mutations as Biomarkers for Metastasis in Colon Cancer
Status: Completed | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Other Study IDs: INST 1204
Record Dates: First submitted 2019-05-08; First posted 2019-05-15 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Either frozen or paraffin embedded colon cancer tissues
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-interventional — Non-interventional

SUMMARY:
This proposal seeks to further understand the contribution of the PIK3CA mutations in colon cancer, by correlating the type of hotspot mutation with the development of metastases in stage II and stage Ill patients.

In order to do this, DNA will be extracted from either frozen or paraffin embedded colon cancer tissues to sequence PIK3CA, KRAS and BRAF. Clinical outcome data will be gathered to include metastases and survival to correlate with PIK3CA, KRAS and BRAF mutational status. Patients with stage II and stage Ill colon cancers will be identified in the University of New Mexico Human Tissue Repository and the NIH PLCO prevention trial biorepository.

Existing banked tissues of stage II and Ill colon cancers will be collected. There will be no direct contact with living individuals. Epidemiological factors such as age, race, gender and outcome data of metastases and survival will be collected.

DETAILED DESCRIPTION:
This proposal aims to identify PIK3CA mutations as a biomarker for metastasis.

In order to do this, DNA will be extracted from either frozen or paraffin embedded colon cancer tissues to sequence PIK3CA, KRAS and BRAF. Clinical outcome data will be gathered to include metastases and survival to correlate with PIK3CA, KRAS and BRAF mutational status. Patients with stage II and stage Ill colon cancers will be identified in the University of New Mexico Human Tissue Repository and the NIH PLCO prevention trial biorepository.

Existing banked tissues of stage II and Ill colon cancers will be collected. There will be no direct contact with living individuals. Epidemiological factors such as age, race, gender and outcome data of metastases and survival will be collected.

Specific Aims:

1. To develop and standardize methods for high throughput DNA extraction and analysis from colon tumors of patients with stage II and stage III disease harboring PIK3CA exon 9 and exon 20 mutations.
2. To determine the correlation between wild type and PIK3CA, PIK3CA exon 9 and PIK3CA exon 20 mutations and development of metastatic disease and overall survival in stage II and stage III patients with colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Specimen from patients with stage II and stage III colon cancer.

Exclusion Criteria:

* Any other stage or type of disease outside of stage II and stage III colon cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specimen from patients with stage II and stage III colon cancer.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2012-05-22 (Actual); Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
The best standardized method for high throughput DNA extraction and analysis from colon tumors of patients | Through study completion, up to 20 years
  Develop and standardize methods for high throughput DNA extraction and analysis from colon tumors of patients with stage II and stage Ill disease harboring PIK3CA exon 9 and exon 20 mutations.
  Currently, commercially available kits to assay for the Pl3K mutations rely on Sanger sequencing of DNA products extracted from formalin fixed paraffin embedded (FFPE) tissues. The presence of a pseudogene on chromosome 22 can interfere with the detection of helical domain mutations. A pyrosequencing technique which allows one to "sequence by synthesis" has been developed to allow the detection of the hotspot PIK3CA mutations without interference from this pseudogene. The investigators propose to modify and expand this pyrosequencing technique to include the additional mutations identified in exons 9 and 20, allowing identifications of nearly 85% of all PIK3CA mutations. Prior to sequencing the investigators will op
The correlation between wild type PIK3CA, PIK3CA exon 9 and PIK3CA exon 20 mutations and developing of metastatic disease and overall colorectal patient survival | Through study completion, up to 20 years
  Tissues from stage II and stage Ill colorectal cancer patients have been identified in the University of New Mexico (UNM) Human Tissue Repository (HTR) and will be available for analysis. Clinical follow up data including the development of metastases, site(s) of metastases and overall survival will be collected from a combination of the tumor registry and the medical records. Additional formalin fixed paraffin embedded tissues from patients with stage II and Ill colorectal cancer will be available from the NCI Prostate, Lung, Colon, Ovary Prevention Trial. Extensive clinical follow-up and survival data are already annotated for patients in this trial and will be available for analysis. Correlation between wild type PIK3CA, exon 9 and exon 20 PIK3CA mutants, KRAS and BRAF mutational status and the occurrence of metastases will be determined. Survival curves will also be generated based on mutational status of the genes listed above.

CONTACTS AND LOCATIONS:
Overall Officials: Ashwani Rajput, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No